CLINICAL TRIAL: NCT02600884
Title: Efficacy Trial of a Brief Parent-Based Adolescent Sexual Health Intervention
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas Health Science Center, Houston (Other)
Responsible Party: Principal Investigator, Diane Santa Maria, Assistant Professor, The University of Texas Health Science Center, Houston
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: HSC-SN-15-0091
Record Dates: First submitted 2015-11-05; First posted 2015-11-09 (Estimated); Last update posted 2023-11-03 (Actual); Status verified 2023-10

CONDITIONS: Increase HPV Vaccination Uptake; Delay Sexual Debut

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Families Talking Together Plus (FTT+HPV) (Experimental): Parents in the experimental group will attend a 1-hour intervention session, receive program materials to use with youth at home, and receive 2 booster phone calls post-intervention. Content of the experimental intervention includes parent-child sexual health communication and HPV vaccination navigation.
  Interventions: Behavioral: Families Talking Together Plus (FTT+HPV)
- Brief motivational interviewing (BMI) (Active Comparator): Parents in the brief motivational interviewing (BMI) group will attend a 1-hour intervention session, receive program materials to use with youth at home, and receive 2 booster phone calls post-intervention. Content of the control intervention includes obesity prevention strategies using motivational interviewing.
  Interventions: Behavioral: Brief motivational interviewing (BMI)

INTERVENTIONS:
Behavioral: Families Talking Together Plus (FTT+HPV) — Intervention parents will attend a 1-hour intervention session and receive program materials to use with youth at home and 2 booster phone calls post intervention. Content of the experimental intervention includes parent child sexual health communication and HPV vaccination navigation.
  Arms: Families Talking Together Plus (FTT+HPV)
Behavioral: Brief motivational interviewing (BMI) — Control parents will attend a 1-hour intervention session and receive program materials to use with youth at home and 2 booster phone calls post intervention. Content of the control intervention includes obesity prevention strategies using motivational interviewing.
  Arms: Brief motivational interviewing (BMI)

SUMMARY:
The purpose of this research study is to evaluate a brief parent-based adolescent sexual health intervention called Families Talking Together Plus (FTT+). FTT+ is based on an established intervention called Families Talking Together (FTT) and will enhance FTT by adding modules on human papillomavirus (HPV). The goal of the study is to evaluate whether FTT will help parents increase sexual health communication, delay adolescent sexual debut, and increase HPV vaccination. FTT will be delivered to parents of minority youth and will be delivered by student nurses.

ELIGIBILITY:
Age limit for parents: minimum = N/A (No limit); maximum = N/A (No limit) Age limit for children: minimum = 11 years; maximum = 14 years

Inclusion Criteria:

* Parent: resides with a child 11-14 years old who attends a participating community center, after-school program, or Boys and Girls Club (BGC)
* Parent: available for a face-to-face or small group session with the PI or student nurse within 2 months of consenting and assenting to participate in the study
* Parent: can read, write, and speak English or Spanish
* Child: between 11-14 years of age

Exclusion Criteria:

* Parent: Without primary custody of child
* Parent: Incarcerated
* Parent: Unable to attend a face-to-face session within 2 months

Min Age: 11 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 1183 (Actual)
Dates: Start 2015-09 (Actual); Primary Completion 2018-11 (Actual); Study Completion 2019-04 (Actual)

PRIMARY OUTCOMES:
Change in parent child communication as assessed by the Families Talking Together Plus HPV (FTT + HPV) survey administered to parents | 1 month
  The FTT + HPV survey is a survey that has been developed by the investigator for this study. The survey is administered at baseline, 1, and 6 months using iPads and is available as Audio Computer-Assisted Self-Interviews in both English and Spanish.
Change in parent child communication as assessed by the FTT + HPV survey administered to parents | 6 months
Change in intentions for sex as assessed by the FTT + HPV survey administered to youths | 1 month
Change in intentions for sex as assessed by the FTT + HPV survey administered to youths | 6 months

SECONDARY OUTCOMES:
Change in parental monitoring as assessed by the FTT + HPV survey administered to parents | 1 month
Change in parental monitoring as assessed by the FTT + HPV survey administered to parents | 6 months
Change in parental involvement as Assessed by the FTT + HPV survey administered to parents | 1 month
Change in parental involvement as assessed by the FTT + HPV survey administered to parents | 6 months
Change in intentions for communication as assessed by the FTT + HPV survey administered to parents | 1 month
Change in intentions for communication as assessed by the FTT + HPV survey administered to parents | 6 months
Change in intentions for HPV vaccination of child as assessed by the FTT + HPV survey administered to parents | 1 month
Change in intentions for HPV vaccination of child as assessed by the FTT + HPV survey administered to parents | 6 months
Change in sexual activity as assessed by the FTT + HPV survey administered to youths | 1 month
Change in sexual activity as assessed by the FTT + HPV survey administered to youths | 6 months
Change in knowledge of HPV risk factors as assessed by the FTT + HPV survey administered to youths | 1 month
Change in knowledge of HPV risk factors as assessed by the FTT + HPV survey administered to youths | 6 months
Change in parental communication as assessed by the FTT + HPV survey administered to youths | 1 month
Change in parental communication as assessed by the FTT + HPV survey administered to youths | 6 months
Change in HPV vaccine received as assessed by the FTT + HPV survey administered to youths | 1 month
Change in HPV vaccine received as assessed by the FTT + HPV survey administered to youths | 6 months

OTHER OUTCOMES:
Change in confidence as sex educators as assessed by the FTT + HPV survey administered to student nurses | 1 month
Change in confidence as sex educators as assessed by the FTT + HPV survey administered to student nurses | 6 months
Change in intentions to endorse HPV vaccination as assessed by the FTT + HPV survey administered to student nurses | 1 month
Change in intentions to endorse HPV vaccination as assessed by the FTT + HPV survey administered to student nurses | 6 months
Change in knowledge of HPV risk factors as assessed by the FTT + HPV survey administered to student nurses | 1 month
Change in knowledge of HPV risk factors as assessed by the FTT + HPV survey administered to student nurses | 6 months
Change in beliefs as assessed by the FTT + HPV survey administered to student nurses | 1 month
Change in beliefs as assessed by the FTT + HPV survey administered to student nurses | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Diane Santa Maria, DrPH, Principal Investigator — The University of Texas Health Science Center, Houston
Locations (1):
- The University of Texas Health Science Center at Houston, Houston, Texas, United States

REFERENCES:
- [Derived] Coleman DC, Frederick A, Cron S, Markham C, Guilamo-Ramos V, Santa Maria D. Impact of preparing nursing students to deliver a parent-based sexual health intervention on attitudes and intentions for sexual health education and parent communication counseling: a mixed methods study. BMC Nurs. 2023 Oct 10;22(1):375. doi: 10.1186/s12912-023-01531-2. PMID 37817237
- [Derived] Santa Maria D, Markham C, Misra SM, Coleman DC, Lyons M, Desormeaux C, Cron S, Guilamo-Ramos V. Effects of a randomized controlled trial of a brief, student-nurse led, parent-based sexual health intervention on parental protective factors and HPV vaccination uptake. BMC Public Health. 2021 Mar 24;21(1):585. doi: 10.1186/s12889-021-10534-0. PMID 33761920

DOCUMENTS (1):
  • Informed Consent Form (2015-11-13): https://cdn.clinicaltrials.gov/large-docs/84/NCT02600884/ICF_000.pdf